CLINICAL TRIAL: NCT01054625
Title: An Open-label, Multi-Center, Phase I/II Trial Investigating the Pharmacokinetic Profile of Zalutumumab, a Human Monoclonal Epidermal Growth Factor Receptor Antibody in Non-curable Patients With SCCHN
Brief Title: Zalutumumab Pharmacokinetics (PK) in Squamous Cell Carcinoma of the Head and Neck (SCCHN)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Genmab (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GEN211
Record Dates: First submitted 2010-01-15; First posted 2010-01-22 (Estimated); Results first posted 2014-01-03 (Estimated); Last update posted 2023-08-03 (Actual); Status verified 2023-08

CONDITIONS: Head and Neck Cancer
Keywords: Squamous Cell Carcinoma of the Head and Neck; Head and Neck Cancer; Head and Neck Neoplasms; anti-EGFr monoclonal antibody; Zalutumumab
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — zalutumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- zalutumumab 4 mg/kg (Experimental): zalutumumab 4 mg/kg iv single infusion week 1,3, 4 and 5
  Interventions: Biological: zalutumumab
- zalutumumab 8 mg/kg (Experimental): zalutumumab 8 mg/kg iv single infusion week 1, 3, 4 and 5
  Interventions: Biological: zalutumumab
- zalutumumab 16 mg/kg (Experimental): zalutumumab 16 mg/kg iv single infusion week 1, 3, 4 and 5
  Interventions: Biological: zalutumumab

INTERVENTIONS:
Biological: zalutumumab — Zalutumumab is a clear to opalescent liquid. It is intended for intravenous infusion following dilution in sterile, pyrogen free, 0.9% NaCl. Patients will be treated at a specified dose of Zalutumumab over a period of 7 weeks. The dose will be 4mg/kg, 8mg/kg or 16mg/kg depending on when they enter the study. The study will begin with 6 patients on 4mg/kg, then 10 patients on 8mg/kg and lastly 10 patients on 16mg/kg.

SUMMARY:
This study is to support current and future Zalutumumab studies by increasing the Pharmacokinetic (PK) knowledge of the drug. PK is the study of how a drug is absorbed (taken up), distributed (moved around), metabolised (broken down) and excreted (removed) by the body, in relation to time. The first PK trial only went up to 8 mg/kg, and, as there has been some indication that the PK profile for the higher and lower doses is different, this needs to be further evaluated. Furthermore, there is a need for more PK data on dosing with 16mg/kg.

The aim with this study is therefore to evaluate the PK profiles at different doses of Zalutumumab and the amount of drug in the blood at different time points after single and multiple doses. The results of this study, combined with data from completed and ongoing Zalutumumab studies, will enable us to provide patients with an effective treatment option which may significantly prolong their survival and/or improve their quality of life.

DETAILED DESCRIPTION:
This study is to look at the Pharmacokinetics (PK) of Zalutumumab in patients with Head and Neck Cancer. 26 participants will be treated with the study drug Zalutumumab at 4 different doses. Zalutumumab will be given at day 0, day 14, day 21 and day 28. Blood samples (for PK and to check the participant's safety) will be taken before drug is given. Blood samples for PK only will be taken directly after drug is given at all treatment visits and also at +3hr and +12hrs on day 0 and day 28 which may require an overnight stay.

Blood samples for PK only are also taken on days between treatments. After treatment on day 28, eight more blood samples will be taken over 3 weeks. On day 49 participants may enter an optional extended treatment period receiving the drug weekly until it is no longer appropriate for the participant (doctor/participant decision or cancer has advanced).

Dosing in the extended treatment period will start at 16mg/kg. The correct dose for the participant will be checked at each visit by looking for the presence and severity of skin rash. This is a common side effect of medicines like Zalutumumab which block the Epidermal Growth Factor Receptor. The severity of the skin rash is used as a guide for dosing. A mild rash could mean more medication is needed, a severe rash will mean the participant needs a break from the medication. End of study is 8 weeks after the last dose of Zalutumumab and blood samples will be taken +4weeks and +8weeks after the last dose of drug.

ELIGIBILITY:
Inclusion Criteria:

* Males and females ≥ 18 years.
* Diagnosis of squamous cell carcinoma of the oral cavity, oropharynx, hypopharynx or larynx, considered incurable with standard therapy. Diagnosis will have been confirmed using a biopsy of the tumour.
* Patients having, based on the investigators judgment, had disease progression and for whom curative therapy is not possible.
* Patients with a WHO performance status ≤ 2 and a life expectancy of greater than 3 months.
* Following receipt of verbal and written information about the study, the patient must provide signed informed consent before any study related activity is carried out.

Exclusion Criteria:

* Patients previously treated with any Epidermal Growth Factor Receptor (EGFR) targeted therapy such as anti-EGFR monoclonal antibodies or small molecule inhibitors within 6 months prior to visit 2 (first treatment).
* Received the following treatments within 4 weeks prior to Visit 2 (first treatment):

  * Cytotoxic or cytostatic anticancer chemotherapy
  * Total tumor resection
  * Radiotherapy of > 50 Gy to gross tumor volume
* Chronic or current infectious disease such as, but not limited to, chronic renal infection, chronic chest infection with bronchiectasis, sinusitis, and tuberculosis
* Clinically significant cardiac disease including unstable angina, acute myocardial infarction within six months from Visit 1 (screening), congestive heart failure, and arrhythmia requiring therapy, with the exception of extra systoles or minor conduction abnormalities
* Significant concurrent, uncontrolled medical condition including, but not limited to, renal, hepatic, haematological, gastrointestinal, endocrine, pulmonary, neurological, cerebral or psychiatric disease
* History of significant cerebrovascular disease
* Known HIV infection
* Known hepatitis B and/or hepatitis C
* Screening laboratory values:

  * Neutrophils < 1.5 x109/l
  * Platelets < 75 x109/l
  * ALAT > 2.5 times the upper limit of normal (unless known liver metastases exceptions will be dealt with on a case by case basis)
  * ALP > 2.5 times the upper limit of normal (unless known liver metastases exceptions will be dealt with on a case by case basis)
  * Bilirubin > 1.5 times the upper limit of normal
  * Creatinine clearance < 50 ml/min (measured or calculated by the CockgroftGault method)
* Patients who have received treatment with any non-marketed drug substance within 4 weeks before Visit 1(screening)
* Current participation in any other interventional clinical study
* Patients with a BMI ≥ 30 kg/m2
* Patients known or suspected of not being able to comply with a study protocol (e.g. due to alcoholism, drug dependency or psychological disorder)
* Breast feeding women or women with a positive pregnancy test at Visit 1 (screening)
* Women of childbearing potential not willing to use adequate contraception such as hormonal birth control or intrauterine device during study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2010-03; Primary Completion 2011-07 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Pascal Machiels, MD, PhD, Principal Investigator — Cliniques Universitaires SaintLuc, Belgium
Locations (7):
- Belgium (2):
  - Cliniques Universitaires SaintLuc, Brussels
  - Uz Leuven - Campus Gasthuisberg, Leuven
- Hungary (2):
  - Uzsoki Hospital, Budapest
  - Vas Megye es Szombathely, Szombathely
- Slovakia (2):
  - Narodny onkologicky ustav, Bratislava
  - FN Tnava, Trnava
- St James's Institute of Oncology, Leeds, United Kingdom

RESULTS

PARTICIPANT FLOW:
Groups:
- Zalutumumab 4 mg/kg: zalutumumab 4 mg/kg iv infusion
- Zalutumumab 8 mg/kg: zalutumumab 8 mg/kg iv infusion
- Zalutumumab 16 mg/kg: zalutumumab 16 mg/kg iv infusion
Period: Overall Study
Arm/Group | Zalutumumab 4 mg/kg | Zalutumumab 8 mg/kg | Zalutumumab 16 mg/kg
Started | 8 (A total of 31 participants were enrolled, 1 participant died before receiving any zalutumumab) | 12 | 10
Completed | 6 | 9 | 9
Not Completed | 2 | 3 | 1

BASELINE CHARACTERISTICS:
Population: Thirty of the 31 enrolled participants were included in the full analysis set (FAS) population. One participant was excluded from the FAS because he died before the first infusion of trial drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Zalutumumab 4 mg/kg | Zalutumumab 8 mg/kg | Zalutumumab 16 mg/kg | Total
Number analyzed (Participants) | 8 | 12 | 10 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 7 | 8 | 21
  >=65 years | 2 | 5 | 2 | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 57 (8) | 63 (11) | 59 (5) | 60 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 0 | 4
  Male | 5 | 11 | 10 | 26
Region of Enrollment [Number; unit: participants]
  Hungary | 1 | 1 | 0 | 2
  Slovakia | 0 | 1 | 3 | 4
  Belgium | 6 | 7 | 6 | 19
  United Kingdom | 1 | 3 | 1 | 5

OUTCOME MEASURES:

1. Primary Outcome: Maximum Plasma Concentration of Zalutumumab After Fourth Infusion
Time Frame: Pre-dose and post dose at multiple timepoints up to end of the study (up to 30 days)
Population: PK parameter calculation for the fourth infusion was not performed for 3 participants: one participant [8 mg/kg] was withdrawn from treatment before infusion 4 and for two participants [4 mg/kg, 8 mg/kg] no infusion 4 was documented and only concentrations before dosing were reported. Overall number of participants analyzed are the number of participants with data available for analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mg/L
Arm/Group | Zalutumumab 4 mg/kg | Zalutumumab 8 mg/kg | Zalutumumab 16 mg/kg
Number analyzed (Participants) | 7 | 10 | 10
mg/L | 104.3 (31) | 258.1 (28) | 494.3 (50)

2. Primary Outcome: Area Under the Curve 0-7 Days
Time Frame: Pre-dose and post dose at multiple timepoints from start of first infusion up to end of last infusion (Day 0 to 7)
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*mg/L
Arm/Group | Zalutumumab 4 mg/kg | Zalutumumab 8 mg/kg | Zalutumumab 16 mg/kg
Number analyzed (Participants) | 7 | 10 | 10
h*mg/L | 9308 (47) | 25091 (36) | 52158 (57)

3. Secondary Outcome: Area Under the Curve 0-21 Days
Time Frame: Pre-dose and post dose at multiple timepoints from start of fourth infusion up to end of last infusion (Day 0 to 21)
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*mg/L
Arm/Group | Zalutumumab 4 mg/kg | Zalutumumab 8 mg/kg | Zalutumumab 16 mg/kg
Number analyzed (Participants) | 7 | 10 | 10
h*mg/L | 12728 (60.9) | 44275 (43.1) | 105960 (58.8)

4. Secondary Outcome: Elimination Half-life
Time Frame: Pre-dose and post dose at multiple timepoints up to end of the study (up to 30 days)
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h
Arm/Group | Zalutumumab 4 mg/kg | Zalutumumab 8 mg/kg | Zalutumumab 16 mg/kg
Number analyzed (Participants) | 7 | 10 | 10
h | 63 (71.7) | 193 (37.7) | 283 (38.0)

5. Secondary Outcome: Clearance
Time Frame: Pre-dose and post dose at multiple timepoints up to end of the study (up to 30 days)
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | Zalutumumab 4 mg/kg | Zalutumumab 8 mg/kg | Zalutumumab 16 mg/kg
Number analyzed (Participants) | 7 | 10 | 10
L/h | 0.025 (56.3) | 0.018 (25.7) | 0.019 (40.6)

6. Secondary Outcome: Apparent Volume of Distribution During the Terminal Phase
Time Frame: Pre-dose and post dose at multiple timepoints up to end of the study (up to 30 days)
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L
Arm/Group | Zalutumumab 4 mg/kg | Zalutumumab 8 mg/kg | Zalutumumab 16 mg/kg
Number analyzed (Participants) | 7 | 10 | 10
L | 2.28 (49) | 4.99 (35) | 7.83 (56)

7. Secondary Outcome: Apparent Volume of Distribution at Steady State
Time Frame: Pre-dose and post dose at multiple timepoints up to end of the study (up to 30 days)
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L
Arm/Group | Zalutumumab 4 mg/kg | Zalutumumab 8 mg/kg | Zalutumumab 16 mg/kg
Number analyzed (Participants) | 7 | 10 | 10
L | 3.23 (27) | 4.86 (29) | 7.72 (60)

ADVERSE EVENTS:
Time Frame: From first dose until the end of the safety follow-up period (30 days after last dose) up to 60 days
Arm/Group | Zalutumumab 4 mg/kg | Zalutumumab 8 mg/kg | Zalutumumab 16 mg/kg
Serious Adverse Events (participants affected / at risk) | 7/8 | 5/12 | 3/10
Other Adverse Events (participants affected / at risk) | 8/8 | 12/12 | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zalutumumab 4 mg/kg (N=8) | Zalutumumab 8 mg/kg (N=12) | Zalutumumab 16 mg/kg (N=10)
Disease progression (General disorders) | 3 (3) | 4 (4) | 3 (3)
Infusion related reaction (General disorders) | 2 (2) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zalutumumab 4 mg/kg (N=8) | Zalutumumab 8 mg/kg (N=12) | Zalutumumab 16 mg/kg (N=10)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 3 (3)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 1 (1) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 3 (3) | 2 (2)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 3 (3) | 1 (1) | 1 (1)
Glossodynia (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 1 (2) | 2 (2)
Oral pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (3)
Chills (General disorders) | 2 (2) | 1 (1) | 0 (0)
Fatigue (General disorders) | 2 (2) | 5 (5) | 2 (2)
Mucosal inflammation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Pyrexia (General disorders) | 2 (3) | 1 (1) | 2 (2)
Infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 3 (3) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 3 (3) | 4 (4) | 2 (2)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 0 (0)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 2 (2)
Dizziness (Nervous system disorders) | 2 (2) | 1 (1) | 2 (2)
Headache (Nervous system disorders) | 0 (0) | 4 (5) | 2 (2)
Agitation (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (4) | 2 (2)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (2) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 6 (8) | 6 (7)
Hypotension (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The site and the PI may be required to withhold the publication for up to 90 days. Subject to a reasoned request from the sponsor, the publication may be further delayed for a period up to 6 months from the date of first submission to the sponsor.

The sponsor has the right to require deletion of any trade secret, proprietary, or confidential information supplied by the sponsor to the site or the PI. The sponsor shall not otherwise have the right to censor publications.